CLINICAL TRIAL: NCT06802406
Title: Nutrition OUtReach In Systems of Healthcare
Acronym: NOURISH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Duke University (Other); Stanford University (Other); Memorial Sloan-Kettering Cancer Center, USA (Unknown); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NOURISH; R01NR021468 (NIH)
Record Dates: First submitted 2024-12-11; First posted 2025-01-31 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION; Autologous Haemopoietic Stem Cell Transplant; CAR-T Cell Therapy; Food Insecurity
Keywords: nutrition, food insecurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information Group (No Intervention): These participants will receive information on their local food banks according to standard of care.
- Food Bags Group (Experimental): Patients will be given bags of shelf-stable food for 2-3 days for one individual twice a week in clinic. Additionally, they will receive recipes, handouts, and videos to help with education and food preparation.
  Interventions: Other: Food Bags

INTERVENTIONS:
Other: Food Bags — Participants will receive bags of shelf-stable food for 2-3 days for one individual twice a week in clinic. They will also receive recipes, handouts, and videos to help with education and food preparation.
  Other Names: NOURISH
  Arms: Food Bags Group

SUMMARY:
Many children and adults receiving medical treatments have higher costs, which can make it harder for them to afford groceries. When someone can't afford enough food, and they do not receive proper nutrition it can make treatment more difficult.

By doing this study investigators hope to learn more about whether addressing food insecurity by giving patients bags of food in clinic can help improve nutrition, reduce costs, and improve transplant and cellular therapy outcomes.

DETAILED DESCRIPTION:
Food insecurity (FI), defined as a lack of consistent access to enough food for every person in a household to live an active, healthy life due to insufficient money or other resources, affects 17 million (12.8%) of American households. FI is exacerbated in patients with complex medical conditions, and it is associated with worse health outcomes and increased healthcare utilization and costs. Strategies to address FI such as home-delivered meals or food assistance programs like the Supplemental Nutrition Assistance Program (SNAP) and food banks/pantries/pharmacies may improve healthcare outcomes. However, home-delivered meals are associated with higher costs due to individualized delivery while food assistance programs have several barriers to participation. We propose to leverage the strengths of both those approaches in a novel healthcare-community partnership between cancer centers and food banks called Nutrition OUtReach In Systems of Healthcare (NOURISH), to directly deliver food to patients in clinic. Patients, caregivers, dietitians, social workers, nurses, physicians, food bank staff, and community members will work together to determine medically tailored options for the patient population; food banks will oversee sourcing and preparing bags of food; and healthcare providers will distribute bags to patients in clinic after their appointments. Because NOURISH does not require patients to make an extra trip and bags are distributed discreetly to avoid stigma, it increases adoption; because food is handed out in clinic, it lowers costs. We propose to evaluate NOURISH in a multicenter randomized controlled trial in FI patients with hematologic malignancies receiving transplant and cellular therapy (TCT). We chose this population for three reasons: (1) TCT patients are in great need as approximately 75% will relocate to live near a quaternary cancer center (QCC) for a month or more while receiving TCT, removing them from their normal sources of support; (2) TCT patients are at high risk for malnutrition and other adverse outcomes, often struggling with nausea, anorexia, and other side effects that can be exacerbated by FI; (3) TCT may be a model for sustaining care: while other Food is Medicine initiatives have shown economic benefits, because cost savings do not flow to healthcare systems, there is little incentive for implementation. In contrast, TCT is among the most expensive medical procedures, and healthcare systems are typically reimbursed through bundled payments. As a result, QCCs have an incentive to pursue strategies that may lower costs and improve outcomes. For example, many TCT patients with FI will receive total parenteral nutrition, at significant cost. NOURISH may prevent malnutrition and the need for intravenous nutrition through much cheaper food assistance. The success of our randomized controlled trial will provide a compelling rationale for QCCs to continue to fund food banks in their communities, providing much-needed financial support to sustain these partnerships while improving access and outcomes for patients. Furthermore, positive experiences in TCT may lead to the expansion of these healthcare-community partnerships to the broader cancer population and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Planning to receive transplant or cell therapy
* Screen positive for food insecurity by answering "often true" or "sometimes true" to one of the following:

  * "Within the past 12 months, you worried that your food would run out before you got money to buy more,"
  * "Within the past 12 months, the food you bought just didn't last and you didn't have money to get more."
* Age 8 - 80
* Able to read/write English or Spanish (many patient-reported outcome measures lack validated translations in other languages)

Exclusion Criteria:

* Patients who do not tolerate oral nutrition at the time of study enrollment

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Peri-Transplant and Cell Therapy Malnutrition | Through Day 100
  Assessed by Global Leader Initiative on Malnutrition and confirmed by a dietitian

SECONDARY OUTCOMES:
Peri-TCT Incidence of Infections | Through Day 100
  Incidence and subtypes (blood stream, respiratory, or other) of infections captured as standard of care.
Peri-TCT Incidence of Acute Graft-vs-Host-Disease | Through Day 180
  Incidence of acute GVHD captured as standard of care.
Peri-TCT Incidence of Chronic Graft-vs-Host Disease | Through Year 1
  Incidence of chronic GVHD captured as standard of care.
Incidence of Relapse | Through Year 1
  Incidence of relapse captured as standard of care.
Incidence of Treatment-Related Mortality | Through End of Study
  Incidence of treatment-related mortality captured as standard of care.
Overall Survival | Through Year 1
  Overall survival captured as standard of care.
Quality of Life (PROMIS-29 Score) | At Day 100 and at Year 1
  Quality of life as measured by Patient-Reported Outcome Measurement Information System-29 (PROMIS-29) score. The PROMIS-29 uses a scale of 1 to 5, with higher numbers representing a higher frequency, intensity, or duration.
Financial Toxicity | Day 100 and Year 1
  Financial toxicity measured by average Functional Assessment in Chronic Illness Therapy-COST: A FACIT Measure of Financial Toxicity (FACIT-COST) score. The FACIT-COST result scale ranges from a minimum of 0 to a maximum of 44, with a higher number representing better financial well-being.
Physical Function | At Day 100 and at Year 1
  Physical function measured by average 6 minute walk test distance.
Cognitive Function | At Day 100 and at Year 1
  Cognitive function measured by average MOntreal Cognitive Assessment (MOCA) score. The MOCA score ranges from a minimum of 0 to a maximum of 30, with a higher score indicating better cognitive function.
Mental Health | At Day 100 and at Year 1
  Mental health as measured by percentage of patients who are positive on the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 uses a scale ranging from a minimum of 0 to a maximum of 27, interpreted as 1-13: mild depression; 14-19: moderate depression; and 20-27: severe depression.
Dietary Habits and Consumption | At Year 1
  Dietary habits and consumption measured by overall diet quality scores assessed using the Healthy Eating Index (HEI)-2020. The HEI-2020 uses a scale ranging from a minimum of 0 to a maximum of 100, with a higher number indicating a diet more closely aligned with recommended dietary guidelines.
Dietary Habits and Consumption | At Year 1
  Dietary habits and consumption measured by overall diet quality scores assessed using the National Cancer Institute (NCI) Multi-Factor Screener. The NCI Multifactor Screener provides an estimate of intake of percent energy from fat consumed per day.
Dietary Habits and Consumption | At Year 1
  Dietary habits and consumption measured by overall diet quality scores assessed using the National Cancer Institute (NCI) Multi-Factor Screener. The NCI Multifactor Screener provides an intake estimate of fiber (grams) consumed per day.
Dietary Habits and Consumption | At Year 1
  Dietary habits and consumption measured by overall diet quality scores assessed using the National Cancer Institute (NCI) Multi-Factor Screener. The NCI Multifactor Screener provides an estimate of fruit and vegetable intake (servings) consumed per day.
Dietary Habits and Consumption | At Year 1
  Dietary habits and consumption measured by overall diet quality scores assessed using the World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) Cancer Prevention Score. The WCRF/AICR Cancer Prevention Score ranges from a minimum of 0 to a maximum of 10, with a higher number representing greater adherence to cancer prevention recommendations.
Impact on Food Insecurity | At Year 1
  Measured by the United States Department of Agriculture Adult Food Security Module (USDA AFSM) Short Form survey. The USDA AFSM Short Form Survey uses a raw scoring scale from a minimum of 0 to a maximum of 6, with a higher number indicating greater food insecurity.
Social Determinants of Health | At workup and at Year 1
  Social determinants of health measured by the Centers for Medicare & Medicaid Services Accountable Health Communities Health Related Social Needs (CMS AHC HRSN)10-item survey tool.
Fried Frailty | At Day 100 and at Year 1
  Fried Frailty measured by percentage of patients meeting 3 or more of the diagnostic criteria for frailty.

OTHER OUTCOMES:
Muscle Health | At Day 100 and at Year 1
  Muscle health as assessed by MuscleSound, which quantifies changes in intramuscular adipose tissue (kg).
Muscle Health | At Day 100 and at Year 1
  Muscle health as assessed by MuscleSound, which quantifies changes in glycogen stores (g).
Muscle Health | At Day 100 and at Year 1
  Muscle health as assessed by MuscleSound, which quantifies changes in muscle wasting using the Skeletal Muscle Index (SMI), with a higher number representing greater muscle mass.
Muscle Health | At Day 100 and at Year 1
  Muscle health as assessed by MuscleSound, which quantifies changes in the presence or absence of sarcopenia.
Accelerated Aging | At Year 1
  Accelerated aging as measured by evaluation of blood biomarkers in plasma and peripheral blood mononuclear cells.
Home Food Bank Utilization | At Year 1
  Home food bank utilization as measured by percentage of patients reporting use of food bank after intervention.
Impact of NOURISH on Reducing Healthcare Costs | At Year 1
  Impact of NOURISH on all-cause medical resource use and associated costs as measured by the Functional Assessment of Chronic Illness Therapy-COST A FACIT Measure of Financial Toxicity (FACIT-COST) score. The FACIT-COST result scale ranges from a minimum of 0 to a maximum of 44, with a higher number representing better financial well-being.
Impact of NOURISH on Reducing Healthcare Costs | At Year 1
  Impact of NOURISH on costs of resources to support the NOURISH intervention as measured by the study budget.
Impact of NOURISH on Reducing Healthcare Costs | At Year 1
  Impact of NOURISH on preference-weighted measure of health status, as measured by the Euro Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L).
Impact on Participant Microbiome | At Year 1
  Impact on participant microbiome as measured by 16S and/or shotgun sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - University of Kansas Cancer Center, Fairway, Kansas
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis DH, Creavin ST, Yip JL, Noel-Storr AH, Brayne C, Cullum S. Montreal Cognitive Assessment for the detection of dementia. Cochrane Database Syst Rev. 2021 Jul 13;7(7):CD010775. doi: 10.1002/14651858.CD010775.pub3. PMID 34255351
- [Background] Schluter J, Peled JU, Taylor BP, Markey KA, Smith M, Taur Y, Niehus R, Staffas A, Dai A, Fontana E, Amoretti LA, Wright RJ, Morjaria S, Fenelus M, Pessin MS, Chao NJ, Lew M, Bohannon L, Bush A, Sung AD, Hohl TM, Perales MA, van den Brink MRM, Xavier JB. The gut microbiota is associated with immune cell dynamics in humans. Nature. 2020 Dec;588(7837):303-307. doi: 10.1038/s41586-020-2971-8. Epub 2020 Nov 25. PMID 33239790
- [Background] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Background] Hussaini SMQ, Ren Y, Racioppi A, Lew MV, Bohannon L, Johnson E, Li Y, Thompson JC, Henshall B, Darby M, Choi T, Lopez RD, Sarantopoulos S, Gasparetto C, Long GD, Horwitz ME, Chao NJ, Zafar SY, Sung AD. Financial Toxicity and Quality of Life in Patients Undergoing Stem-Cell Transplant Evaluation: A Single-Center Analysis. JCO Oncol Pract. 2024 Mar;20(3):351-360. doi: 10.1200/OP.23.00243. Epub 2023 Dec 21. PMID 38127876
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Clinton SK, Giovannucci EL, Hursting SD. The World Cancer Research Fund/American Institute for Cancer Research Third Expert Report on Diet, Nutrition, Physical Activity, and Cancer: Impact and Future Directions. J Nutr. 2020 Apr 1;150(4):663-671. doi: 10.1093/jn/nxz268. PMID 31758189
- [Background] Shams-White MM, Romaguera D, Mitrou P, Reedy J, Bender A, Brockton NT. Further Guidance in Implementing the Standardized 2018 World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) Score. Cancer Epidemiol Biomarkers Prev. 2020 May;29(5):889-894. doi: 10.1158/1055-9965.EPI-19-1444. Epub 2020 Mar 9. PMID 32152215
- [Background] Shams-White MM, Brockton NT, Mitrou P, Romaguera D, Brown S, Bender A, Kahle LL, Reedy J. Operationalizing the 2018 World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) Cancer Prevention Recommendations: A Standardized Scoring System. Nutrients. 2019 Jul 12;11(7):1572. doi: 10.3390/nu11071572. PMID 31336836
- [Background] David LA, Weil A, Ryan ET, Calderwood SB, Harris JB, Chowdhury F, Begum Y, Qadri F, LaRocque RC, Turnbaugh PJ. Gut microbial succession follows acute secretory diarrhea in humans. mBio. 2015 May 19;6(3):e00381-15. doi: 10.1128/mBio.00381-15. PMID 25991682
- [Background] Siamakpour-Reihani S, Cao F, Lyu J, Ren Y, Nixon AB, Xie J, Bush AT, Starr MD, Bain JR, Muehlbauer MJ, Ilkayeva O, Byers Kraus V, Huebner JL, Chao NJ, Sung AD. Evaluating immune response and metabolic related biomarkers pre-allogenic hematopoietic stem cell transplant in acute myeloid leukemia. PLoS One. 2022 Jun 14;17(6):e0268963. doi: 10.1371/journal.pone.0268963. eCollection 2022. PMID 35700185
- [Background] Parker D, Sloane R, Pieper CF, Hall KS, Kraus VB, Kraus WE, Huebner JL, Ilkayeva OR, Bain JR, Newby LK, Cohen HJ, Morey MC. Age-Related Adverse Inflammatory and Metabolic Changes Begin Early in Adulthood. J Gerontol A Biol Sci Med Sci. 2019 Feb 15;74(3):283-289. doi: 10.1093/gerona/gly121. PMID 29985987
- [Background] Maecker HT, McCoy JP, Nussenblatt R. Standardizing immunophenotyping for the Human Immunology Project. Nat Rev Immunol. 2012 Feb 17;12(3):191-200. doi: 10.1038/nri3158. PMID 22343568
- [Background] Alsaggaf R, Katta S, Wang T, Hicks BD, Zhu B, Spellman SR, Lee SJ, Horvath S, Gadalla SM. Epigenetic Aging and Hematopoietic Cell Transplantation in Patients With Severe Aplastic Anemia. Transplant Cell Ther. 2021 Apr;27(4):313.e1-313.e8. doi: 10.1016/j.jtct.2021.01.013. Epub 2021 Jan 16. PMID 33836872
- [Background] Ulrich S, Hildenbrand FF, Treder U, Fischler M, Keusch S, Speich R, Fasnacht M. Reference values for the 6-minute walk test in healthy children and adolescents in Switzerland. BMC Pulm Med. 2013 Aug 5;13:49. doi: 10.1186/1471-2466-13-49. PMID 23915140
- [Background] Rudolphi JM, Berg RL. Mental health of agricultural adolescents and adults: Preliminary results of a five-year study. Front Public Health. 2023 Mar 2;11:1056487. doi: 10.3389/fpubh.2023.1056487. eCollection 2023. PMID 36935670
- [Background] Pike NA, Poulsen MK, Woo MA. Validity of the Montreal Cognitive Assessment Screener in Adolescents and Young Adults With and Without Congenital Heart Disease. Nurs Res. 2017 May/Jun;66(3):222-230. doi: 10.1097/NNR.0000000000000192. PMID 28448372
- [Background] Kreimeier S, Astrom M, Burstrom K, Egmar AC, Gusi N, Herdman M, Kind P, Perez-Sousa MA, Greiner W. EQ-5D-Y-5L: developing a revised EQ-5D-Y with increased response categories. Qual Life Res. 2019 Jul;28(7):1951-1961. doi: 10.1007/s11136-019-02115-x. Epub 2019 Feb 9. PMID 30739287
- [Background] DeWalt DA, Gross HE, Gipson DS, Selewski DT, DeWitt EM, Dampier CD, Hinds PS, Huang IC, Thissen D, Varni JW. PROMIS((R)) pediatric self-report scales distinguish subgroups of children within and across six common pediatric chronic health conditions. Qual Life Res. 2015 Sep;24(9):2195-208. doi: 10.1007/s11136-015-0953-3. Epub 2015 Feb 26. PMID 25715946
- [Background] Dee EC. Family and Caregiver Financial Toxicity Associated With Cancer-A Global, Inequitable, and Urgent Consideration. JAMA Netw Open. 2023 Jun 1;6(6):e2319317. doi: 10.1001/jamanetworkopen.2023.19317. No abstract available. PMID 37347488
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Petrone BL, Aqeel A, Jiang S, Durand HK, Dallow EP, McCann JR, Dressman HK, Hu Z, Tenekjian CB, Yancy WS Jr, Lin PH, Scialla JJ, Seed PC, Rawls JF, Armstrong SC, Stevens J, David LA. Diversity of plant DNA in stool is linked to dietary quality, age, and household income. Proc Natl Acad Sci U S A. 2023 Jul 4;120(27):e2304441120. doi: 10.1073/pnas.2304441120. Epub 2023 Jun 27. PMID 37368926
- [Background] Young HJ, Jenkins NT, Zhao Q, Mccully KK. Measurement of intramuscular fat by muscle echo intensity. Muscle Nerve. 2015 Dec;52(6):963-71. doi: 10.1002/mus.24656. Epub 2015 Sep 7. PMID 25787260
- [Background] Reimers K, Reimers CD, Wagner S, Paetzke I, Pongratz DE. Skeletal muscle sonography: a correlative study of echogenicity and morphology. J Ultrasound Med. 1993 Feb;12(2):73-7. doi: 10.7863/jum.1993.12.2.73. PMID 8468739
- [Background] Burton AM, Stock MS. Consistency of novel ultrasound equations for estimating percent intramuscular fat. Clin Physiol Funct Imaging. 2018 Jun 11. doi: 10.1111/cpf.12532. Online ahead of print. PMID 29888525
- [Background] Tsuruta Y, Rogers LQ, Krontiras H, Grizzle WE, Fruge AD, Oster RA, Umphrey HR, Jones LW, Azrad M, Demark-Wahnefried W. Exploring effects of presurgical weight loss among women with stage 0-II breast cancer: protocol for a randomised controlled feasibility trial. BMJ Open. 2016 Sep 15;6(9):e012320. doi: 10.1136/bmjopen-2016-012320. PMID 27633639
- [Background] Pekmezi DW, Crane TE, Oster RA, Rogers LQ, Hoenemeyer T, Farrell D, Cole WW, Wolin K, Badr H, Demark-Wahnefried W. Rationale and Methods for a Randomized Controlled Trial of a Dyadic, Web-Based, Weight Loss Intervention among Cancer Survivors and Partners: The DUET Study. Nutrients. 2021 Sep 29;13(10):3472. doi: 10.3390/nu13103472. PMID 34684474
- [Background] Pekmezi D, Fontaine K, Rogers LQ, Pisu M, Martin MY, Schoenberger-Godwin YM, Oster RA, Kenzik K, Ivankova NV, Demark-Wahnefried W. Adapting MultiPLe behavior Interventions that eFfectively Improve (AMPLIFI) cancer survivor health: program project protocols for remote lifestyle intervention and assessment in 3 inter-related randomized controlled trials among survivors of obesity-related cancers. BMC Cancer. 2022 Apr 29;22(1):471. doi: 10.1186/s12885-022-09519-y. PMID 35488238
- [Background] Demark-Wahnefried W, Jones LW, Snyder DC, Sloane RJ, Kimmick GG, Hughes DC, Badr HJ, Miller PE, Burke LE, Lipkus IM. Daughters and Mothers Against Breast Cancer (DAMES): main outcomes of a randomized controlled trial of weight loss in overweight mothers with breast cancer and their overweight daughters. Cancer. 2014 Aug 15;120(16):2522-34. doi: 10.1002/cncr.28761. Epub 2014 May 7. PMID 24804802
- [Background] Demark-Wahnefried W, Nix JW, Hunter GR, Rais-Bahrami S, Desmond RA, Chacko B, Morrow CD, Azrad M, Fruge AD, Tsuruta Y, Ptacek T, Tully SA, Segal R, Grizzle WE. Feasibility outcomes of a presurgical randomized controlled trial exploring the impact of caloric restriction and increased physical activity versus a wait-list control on tumor characteristics and circulating biomarkers in men electing prostatectomy for prostate cancer. BMC Cancer. 2016 Feb 5;16:61. doi: 10.1186/s12885-016-2075-x. PMID 26850040
- [Background] Conway JM, Ingwersen LA, Vinyard BT, Moshfegh AJ. Effectiveness of the US Department of Agriculture 5-step multiple-pass method in assessing food intake in obese and nonobese women. Am J Clin Nutr. 2003 May;77(5):1171-8. doi: 10.1093/ajcn/77.5.1171. PMID 12716668
- [Background] Conway JM, Ingwersen LA, Moshfegh AJ. Accuracy of dietary recall using the USDA five-step multiple-pass method in men: an observational validation study. J Am Diet Assoc. 2004 Apr;104(4):595-603. doi: 10.1016/j.jada.2004.01.007. PMID 15054345
- [Background] Freedman LS, Commins JM, Willett W, Tinker LF, Spiegelman D, Rhodes D, Potischman N, Neuhouser ML, Moshfegh AJ, Kipnis V, Baer DJ, Arab L, Prentice RL, Subar AF. Evaluation of the 24-Hour Recall as a Reference Instrument for Calibrating Other Self-Report Instruments in Nutritional Cohort Studies: Evidence From the Validation Studies Pooling Project. Am J Epidemiol. 2017 Jul 1;186(1):73-82. doi: 10.1093/aje/kwx039. PMID 28402488
- [Background] Yin L, Lin X, Zhao Z, Li N, He X, Zhang M, Yang J, Guo Z, Li Z, Wang K, Weng M, Cong M, Li S, Li T, Ma H, Ba Y, Li W, Cui J, Liu J, Song C, Shi H, Xu H. Is hand grip strength a necessary supportive index in the phenotypic criteria of the GLIM-based diagnosis of malnutrition in patients with cancer? Support Care Cancer. 2021 Jul;29(7):4001-4013. doi: 10.1007/s00520-020-05975-z. Epub 2021 Jan 4. PMID 33398429
- [Background] Jensen GL, Cederholm T, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, de Baptista GA, Barazzoni R, Blaauw R, Coats AJS, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren M, Siltharm S, Singer P, Tappenden KA, Velasco N, Waitzberg DL, Yamwong P, Yu J, Compher C, Van Gossum A. GLIM Criteria for the Diagnosis of Malnutrition: A Consensus Report From the Global Clinical Nutrition Community. JPEN J Parenter Enteral Nutr. 2019 Jan;43(1):32-40. doi: 10.1002/jpen.1440. Epub 2018 Sep 2. PMID 30175461
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Jim HS, Syrjala KL, Rizzo D. Supportive care of hematopoietic cell transplant patients. Biol Blood Marrow Transplant. 2012 Jan;18(1 Suppl):S12-6. doi: 10.1016/j.bbmt.2011.10.029. PMID 22226095
- [Background] Smith PJ, Lew M, Lowder Y, Romero K, Thompson JC, Bohannon L, Pittman A, Artica A, Ramalingam S, Choi T, Gasparetto C, Horwitz M, Long G, Lopez R, Rizzieri D, Sarantopoulos S, Sullivan K, Chao N, Sung AD. Cognitive impairment in candidates for allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2022 Jan;57(1):89-94. doi: 10.1038/s41409-021-01470-z. Epub 2021 Oct 19. PMID 34667271
- [Background] Kang JM, Cho YS, Park S, Lee BH, Sohn BK, Choi CH, Choi JS, Jeong HY, Cho SJ, Lee JH, Lee JY. Montreal cognitive assessment reflects cognitive reserve. BMC Geriatr. 2018 Oct 30;18(1):261. doi: 10.1186/s12877-018-0951-8. PMID 30376815
- [Background] van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value Health. 2012 Jul-Aug;15(5):708-15. doi: 10.1016/j.jval.2012.02.008. Epub 2012 May 24. PMID 22867780
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Aghdaee M, Gu Y, Sinha K, Parkinson B, Sharma R, Cutler H. Mapping the Patient-Reported Outcomes Measurement Information System (PROMIS-29) to EQ-5D-5L. Pharmacoeconomics. 2023 Feb;41(2):187-198. doi: 10.1007/s40273-022-01157-3. Epub 2022 Nov 7. PMID 36336773
- [Background] Engel MD, Shelnutt KP, House LA, El Zein A, Mathews AE. Differences in Measured and Self-Categorized Food Security Status and Related Coping Strategies among College Students. Nutrients. 2022 Aug 30;14(17):3569. doi: 10.3390/nu14173569. PMID 36079826
- [Background] Gibson CJ, Lindsley RC, Tchekmedyian V, Mar BG, Shi J, Jaiswal S, Bosworth A, Francisco L, He J, Bansal A, Morgan EA, Lacasce AS, Freedman AS, Fisher DC, Jacobsen E, Armand P, Alyea EP, Koreth J, Ho V, Soiffer RJ, Antin JH, Ritz J, Nikiforow S, Forman SJ, Michor F, Neuberg D, Bhatia R, Bhatia S, Ebert BL. Clonal Hematopoiesis Associated With Adverse Outcomes After Autologous Stem-Cell Transplantation for Lymphoma. J Clin Oncol. 2017 May 10;35(14):1598-1605. doi: 10.1200/JCO.2016.71.6712. Epub 2017 Jan 9. PMID 28068180
- [Background] Gibson CJ, Kim HT, Zhao L, Murdock HM, Hambley B, Ogata A, Madero-Marroquin R, Wang S, Green L, Fleharty M, Dougan T, Cheng CA, Blumenstiel B, Cibulskis C, Tsuji J, Duran M, Gocke CD, Antin JH, Nikiforow S, DeZern AE, Chen YB, Ho VT, Jones RJ, Lennon NJ, Walt DR, Ritz J, Soiffer RJ, Gondek LP, Lindsley RC. Donor Clonal Hematopoiesis and Recipient Outcomes After Transplantation. J Clin Oncol. 2022 Jan 10;40(2):189-201. doi: 10.1200/JCO.21.02286. Epub 2021 Nov 18. PMID 34793200
- [Background] Fall-Dickson JM, Pavletic SZ, Mays JW, Schubert MM. Oral Complications of Chronic Graft-Versus-Host Disease. J Natl Cancer Inst Monogr. 2019 Aug 1;2019(53):lgz007. doi: 10.1093/jncimonographs/lgz007. PMID 31425593
- [Background] Garios RS, Oliveira PM, Aguiar AS, Luquetti SCPD. Caloric and protein intake in different periods of hospitalization of patients undergoing hematopoietic stem cell transplantation. Hematol Transfus Cell Ther. 2018 Oct-Dec;40(4):332-338. doi: 10.1016/j.htct.2018.02.003. Epub 2018 Apr 18. PMID 30370411
- [Background] Robin M, Porcher R, Ades L, Boissel N, Raffoux E, Xhaard A, Larghero J, Gardin C, Himberlin C, Delmer A, Fenaux P, Dombret H, Socie G, Peffault de Latour R. Matched unrelated or matched sibling donors result in comparable outcomes after non-myeloablative HSCT in patients with AML or MDS. Bone Marrow Transplant. 2013 Oct;48(10):1296-301. doi: 10.1038/bmt.2013.50. Epub 2013 Apr 15. PMID 23584440
- [Background] Horan JT, Logan BR, Agovi-Johnson MA, Lazarus HM, Bacigalupo AA, Ballen KK, Bredeson CN, Carabasi MH, Gupta V, Hale GA, Khoury HJ, Juckett MB, Litzow MR, Martino R, McCarthy PL, Smith FO, Rizzo JD, Pasquini MC. Reducing the risk for transplantation-related mortality after allogeneic hematopoietic cell transplantation: how much progress has been made? J Clin Oncol. 2011 Mar 1;29(7):805-13. doi: 10.1200/JCO.2010.32.5001. Epub 2011 Jan 10. PMID 21220593
- [Background] Gooley TA, Chien JW, Pergam SA, Hingorani S, Sorror ML, Boeckh M, Martin PJ, Sandmaier BM, Marr KA, Appelbaum FR, Storb R, McDonald GB. Reduced mortality after allogeneic hematopoietic-cell transplantation. N Engl J Med. 2010 Nov 25;363(22):2091-101. doi: 10.1056/NEJMoa1004383. PMID 21105791
- [Background] Muscaritoli M, Lucia S, Farcomeni A, Lorusso V, Saracino V, Barone C, Plastino F, Gori S, Magarotto R, Carteni G, Chiurazzi B, Pavese I, Marchetti L, Zagonel V, Bergo E, Tonini G, Imperatori M, Iacono C, Maiorana L, Pinto C, Rubino D, Cavanna L, Di Cicilia R, Gamucci T, Quadrini S, Palazzo S, Minardi S, Merlano M, Colucci G, Marchetti P; PreMiO Study Group. Prevalence of malnutrition in patients at first medical oncology visit: the PreMiO study. Oncotarget. 2017 Aug 10;8(45):79884-79896. doi: 10.18632/oncotarget.20168. eCollection 2017 Oct 3. PMID 29108370
- [Background] Raber M, Jackson A, Basen-Engquist K, Bradley C, Chambers S, Gany FM, Halbert CH, Lindau ST, Perez-Escamilla R, Seligman H. Food Insecurity Among People With Cancer: Nutritional Needs as an Essential Component of Care. J Natl Cancer Inst. 2022 Dec 8;114(12):1577-1583. doi: 10.1093/jnci/djac135. PMID 36130287
- [Background] Patel KG, Borno HT, Seligman HK. Food insecurity screening: A missing piece in cancer management. Cancer. 2019 Oct 15;125(20):3494-3501. doi: 10.1002/cncr.32291. Epub 2019 Jul 9. No abstract available. PMID 31287159
- [Background] Hanson KL, Connor LM. Food insecurity and dietary quality in US adults and children: a systematic review. Am J Clin Nutr. 2014 Aug;100(2):684-92. doi: 10.3945/ajcn.114.084525. Epub 2014 Jun 18. PMID 24944059
- [Background] Silverman J, Krieger J, Kiefer M, Hebert P, Robinson J, Nelson K. The Relationship Between Food Insecurity and Depression, Diabetes Distress and Medication Adherence Among Low-Income Patients with Poorly-Controlled Diabetes. J Gen Intern Med. 2015 Oct;30(10):1476-80. doi: 10.1007/s11606-015-3351-1. Epub 2015 Apr 28. PMID 25917659
- [Background] Gundersen C, Ziliak JP. Food Insecurity And Health Outcomes. Health Aff (Millwood). 2015 Nov;34(11):1830-9. doi: 10.1377/hlthaff.2015.0645. PMID 26526240
- [Background] Reeder N, Tolar-Peterson T, Bailey RH, Cheng WH, Evans MW Jr. Food Insecurity and Depression among US Adults: NHANES 2005-2016. Nutrients. 2022 Jul 27;14(15):3081. doi: 10.3390/nu14153081. PMID 35956257
- [Background] Zenk SN, Tabak LA, Perez-Stable EJ. Research Opportunities to Address Nutrition Insecurity and Disparities. JAMA. 2022 May 24;327(20):1953-1954. doi: 10.1001/jama.2022.7159. No abstract available. PMID 35486390
- [Background] Afulani P, Herman D, Coleman-Jensen A, Harrison GG. Food Insecurity and Health Outcomes Among Older Adults: The Role of Cost-Related Medication Underuse. J Nutr Gerontol Geriatr. 2015;34(3):319-42. doi: 10.1080/21551197.2015.1054575. PMID 26267444
- [Background] Holmes ZC, Tang H, Liu C, Bush A, Neubert BC, Jiao Y, Covington M, Cardona DM, Kirtley MC, Chen BJ, Chao NJ, David LA, Sung AD. Prebiotic galactooligosaccharides interact with mouse gut microbiota to attenuate acute graft-versus-host disease. Blood. 2022 Nov 24;140(21):2300-2304. doi: 10.1182/blood.2021015178. PMID 35930748
- [Background] Thaiss CA, Zmora N, Levy M, Elinav E. The microbiome and innate immunity. Nature. 2016 Jul 7;535(7610):65-74. doi: 10.1038/nature18847. PMID 27383981
- [Background] Honda K, Littman DR. The microbiota in adaptive immune homeostasis and disease. Nature. 2016 Jul 7;535(7610):75-84. doi: 10.1038/nature18848. PMID 27383982
- [Background] Mager LF, Burkhard R, Pett N, Cooke NCA, Brown K, Ramay H, Paik S, Stagg J, Groves RA, Gallo M, Lewis IA, Geuking MB, McCoy KD. Microbiome-derived inosine modulates response to checkpoint inhibitor immunotherapy. Science. 2020 Sep 18;369(6510):1481-1489. doi: 10.1126/science.abc3421. Epub 2020 Aug 13. PMID 32792462
- [Background] Zheng L, Kelly CJ, Battista KD, Schaefer R, Lanis JM, Alexeev EE, Wang RX, Onyiah JC, Kominsky DJ, Colgan SP. Microbial-Derived Butyrate Promotes Epithelial Barrier Function through IL-10 Receptor-Dependent Repression of Claudin-2. J Immunol. 2017 Oct 15;199(8):2976-2984. doi: 10.4049/jimmunol.1700105. Epub 2017 Sep 11. PMID 28893958
- [Background] Kelly CJ, Zheng L, Campbell EL, Saeedi B, Scholz CC, Bayless AJ, Wilson KE, Glover LE, Kominsky DJ, Magnuson A, Weir TL, Ehrentraut SF, Pickel C, Kuhn KA, Lanis JM, Nguyen V, Taylor CT, Colgan SP. Crosstalk between Microbiota-Derived Short-Chain Fatty Acids and Intestinal Epithelial HIF Augments Tissue Barrier Function. Cell Host Microbe. 2015 May 13;17(5):662-71. doi: 10.1016/j.chom.2015.03.005. Epub 2015 Apr 9. PMID 25865369
- [Background] Metzger KE, Rucker Y, Callaghan M, Churchill M, Jovanovic BD, Zembower TR, Bolon MK. The burden of mucosal barrier injury laboratory-confirmed bloodstream infection among hematology, oncology, and stem cell transplant patients. Infect Control Hosp Epidemiol. 2015 Feb;36(2):119-24. doi: 10.1017/ice.2014.38. PMID 25632993
- [Background] Dandoy CE, Kim S, Chen M, Ahn KW, Ardura MI, Brown V, Chhabra S, Diaz MA, Dvorak C, Farhadfar N, Flagg A, Ganguly S, Hale GA, Hashmi SK, Hematti P, Martino R, Nishihori T, Nusrat R, Olsson RF, Rotz SJ, Sung AD, Perales MA, Lindemans CA, Komanduri KV, Riches ML. Incidence, Risk Factors, and Outcomes of Patients Who Develop Mucosal Barrier Injury-Laboratory Confirmed Bloodstream Infections in the First 100 Days After Allogeneic Hematopoietic Stem Cell Transplant. JAMA Netw Open. 2020 Jan 3;3(1):e1918668. doi: 10.1001/jamanetworkopen.2019.18668. PMID 31913492
- [Background] Sung AD, Chao NJ. Concise review: acute graft-versus-host disease: immunobiology, prevention, and treatment. Stem Cells Transl Med. 2013 Jan;2(1):25-32. doi: 10.5966/sctm.2012-0115. Epub 2012 Dec 19. PMID 23283494
- [Background] Campbell SC, Wisniewski PJ, Noji M, McGuinness LR, Haggblom MM, Lightfoot SA, Joseph LB, Kerkhof LJ. The Effect of Diet and Exercise on Intestinal Integrity and Microbial Diversity in Mice. PLoS One. 2016 Mar 8;11(3):e0150502. doi: 10.1371/journal.pone.0150502. eCollection 2016. PMID 26954359
- [Background] Bressa C, Bailen-Andrino M, Perez-Santiago J, Gonzalez-Soltero R, Perez M, Montalvo-Lominchar MG, Mate-Munoz JL, Dominguez R, Moreno D, Larrosa M. Differences in gut microbiota profile between women with active lifestyle and sedentary women. PLoS One. 2017 Feb 10;12(2):e0171352. doi: 10.1371/journal.pone.0171352. eCollection 2017. PMID 28187199
- [Background] Evans CC, LePard KJ, Kwak JW, Stancukas MC, Laskowski S, Dougherty J, Moulton L, Glawe A, Wang Y, Leone V, Antonopoulos DA, Smith D, Chang EB, Ciancio MJ. Exercise prevents weight gain and alters the gut microbiota in a mouse model of high fat diet-induced obesity. PLoS One. 2014 Mar 26;9(3):e92193. doi: 10.1371/journal.pone.0092193. eCollection 2014. PMID 24670791
- [Background] Denou E, Marcinko K, Surette MG, Steinberg GR, Schertzer JD. High-intensity exercise training increases the diversity and metabolic capacity of the mouse distal gut microbiota during diet-induced obesity. Am J Physiol Endocrinol Metab. 2016 Jun 1;310(11):E982-93. doi: 10.1152/ajpendo.00537.2015. Epub 2016 Apr 26. PMID 27117007
- [Background] Stein-Thoeringer CK, Nichols KB, Lazrak A, Docampo MD, Slingerland AE, Slingerland JB, Clurman AG, Armijo G, Gomes ALC, Shono Y, Staffas A, Burgos da Silva M, Devlin SM, Markey KA, Bajic D, Pinedo R, Tsakmaklis A, Littmann ER, Pastore A, Taur Y, Monette S, Arcila ME, Pickard AJ, Maloy M, Wright RJ, Amoretti LA, Fontana E, Pham D, Jamal MA, Weber D, Sung AD, Hashimoto D, Scheid C, Xavier JB, Messina JA, Romero K, Lew M, Bush A, Bohannon L, Hayasaka K, Hasegawa Y, Vehreschild MJGT, Cross JR, Ponce DM, Perales MA, Giralt SA, Jenq RR, Teshima T, Holler E, Chao NJ, Pamer EG, Peled JU, van den Brink MRM. Lactose drives Enterococcus expansion to promote graft-versus-host disease. Science. 2019 Nov 29;366(6469):1143-1149. doi: 10.1126/science.aax3760. PMID 31780560
- [Background] Peled JU, Gomes ALC, Devlin SM, Littmann ER, Taur Y, Sung AD, Weber D, Hashimoto D, Slingerland AE, Slingerland JB, Maloy M, Clurman AG, Stein-Thoeringer CK, Markey KA, Docampo MD, Burgos da Silva M, Khan N, Gessner A, Messina JA, Romero K, Lew MV, Bush A, Bohannon L, Brereton DG, Fontana E, Amoretti LA, Wright RJ, Armijo GK, Shono Y, Sanchez-Escamilla M, Castillo Flores N, Alarcon Tomas A, Lin RJ, Yanez San Segundo L, Shah GL, Cho C, Scordo M, Politikos I, Hayasaka K, Hasegawa Y, Gyurkocza B, Ponce DM, Barker JN, Perales MA, Giralt SA, Jenq RR, Teshima T, Chao NJ, Holler E, Xavier JB, Pamer EG, van den Brink MRM. Microbiota as Predictor of Mortality in Allogeneic Hematopoietic-Cell Transplantation. N Engl J Med. 2020 Feb 27;382(9):822-834. doi: 10.1056/NEJMoa1900623. PMID 32101664
- [Background] Khan N, Lindner S, Gomes ALC, Devlin SM, Shah GL, Sung AD, Sauter CS, Landau HJ, Dahi PB, Perales MA, Chung DJ, Lesokhin AM, Dai A, Clurman A, Slingerland JB, Slingerland AE, Brereton DG, Giardina PA, Maloy M, Armijo GK, Rondon-Clavo C, Fontana E, Bohannon L, Ramalingam S, Bush AT, Lew MV, Messina JA, Littmann E, Taur Y, Jenq RR, Chao NJ, Giralt S, Markey KA, Pamer EG, van den Brink MRM, Peled JU. Fecal microbiota diversity disruption and clinical outcomes after auto-HCT: a multicenter observational study. Blood. 2021 Mar 18;137(11):1527-1537. doi: 10.1182/blood.2020006923. PMID 33512409
- [Background] Guo H, Chou WC, Lai Y, Liang K, Tam JW, Brickey WJ, Chen L, Montgomery ND, Li X, Bohannon LM, Sung AD, Chao NJ, Peled JU, Gomes ALC, van den Brink MRM, French MJ, Macintyre AN, Sempowski GD, Tan X, Sartor RB, Lu K, Ting JPY. Multi-omics analyses of radiation survivors identify radioprotective microbes and metabolites. Science. 2020 Oct 30;370(6516):eaay9097. doi: 10.1126/science.aay9097. PMID 33122357
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Bieniek J, Wilczynski K, Szewieczek J. Fried frailty phenotype assessment components as applied to geriatric inpatients. Clin Interv Aging. 2016 Apr 22;11:453-9. doi: 10.2147/CIA.S101369. eCollection 2016. PMID 27217729
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] de Souza JA, Yap BJ, Hlubocky FJ, Wroblewski K, Ratain MJ, Cella D, Daugherty CK. The development of a financial toxicity patient-reported outcome in cancer: The COST measure. Cancer. 2014 Oct 15;120(20):3245-53. doi: 10.1002/cncr.28814. Epub 2014 Jun 20. PMID 24954526
- [Background] Billioux A, Conway PH, Alley DE. Addressing Population Health: Integrators in the Accountable Health Communities Model. JAMA. 2017 Nov 21;318(19):1865-1866. doi: 10.1001/jama.2017.15063. No abstract available. PMID 29049552
- [Background] Alley DE, Asomugha CN, Conway PH, Sanghavi DM. Accountable Health Communities--Addressing Social Needs through Medicare and Medicaid. N Engl J Med. 2016 Jan 7;374(1):8-11. doi: 10.1056/NEJMp1512532. Epub 2016 Jan 5. No abstract available. PMID 26731305
- [Background] Lew MV, Ren Y, Lowder YP, Siamakpour-Reihani S, Ramalingam S, Romero KM, Thompson JC, Bohannon LM, McIntyre J, Tang H, Van Opstal J, Johnson E, Cohen HJ, Bartlett DB, Pastva AM, Morey M, Hall KS, Smith P, Peters KB, Somers TJ, Kelleher S, Smith SK, Wischmeyer PE, Lin PH, Wood WA, Thorpe G, Minor K, Wiggins K, Hennig T, Helms T, Welch R, Matthews B, Liu J, Burleson J, Aberant T, Engemann AK, Henshall B, Darby M, Proch C, Dellascio M, Pittman A, Suminguit J, Choi T, Gasparetto C, Long GD, Lopez RD, Sarantopoulos S, Horwitz ME, Chao NJ, Sung AD. Geriatric Assessment Reveals Actionable Impairments in Hematopoietic Stem Cell Transplantation Candidates Age 18 to 80 Years. Transplant Cell Ther. 2022 Aug;28(8):498.e1-498.e9. doi: 10.1016/j.jtct.2022.05.018. Epub 2022 May 17. PMID 35595226
- [Background] Broder MS, Quock TP, Chang E, Reddy SR, Agarwal-Hashmi R, Arai S, Villa KF. The Cost of Hematopoietic Stem-Cell Transplantation in the United States. Am Health Drug Benefits. 2017 Oct;10(7):366-374. PMID 29263771
- See also: Healthy People 2030 - Food Insecurity — https://health.gov/healthypeople/priority-areas/social-determinants-health/literature-summaries/food-insecurity
- See also: The Impact Of Food Insecurity On Adult Health & Well-Being — https://healthcare.rti.org/insights/food-insecurity-adult-health
- See also: What are the implications of food insecurity for health and health care? — https://proof.utoronto.ca/food-insecurity/what-are-the-implications-of-food-insecurity-for-health-and-health-care/
- See also: Compromises and Coping Strategies 2014 — https://www.feedingamerica.org/hunger-in-america/impact-of-hunger
- See also: The Impact of Poverty, Food Insecurity, and Poor Nutrition on Health and Well-Being — https://frac.org/wp-content/uploads/hunger-health-impact-poverty-food-insecurity-health-well-being.pdf